CLINICAL TRIAL: NCT05459064
Title: Retrospective Data Collection on the Use of Motiva Flora TE in Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Establishment Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: CLINP-001013
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Motiva Flora TE — This is a retrospective, observational study - collecting data on patients who have gone through the staged procedure with the Motiva Flora Tissue Expander / Long-term breast implant.

SUMMARY:
The Motiva Flora® TE are intended for temporary subcutaneous or submuscular implantation to develop surgical flaps and additional tissue coverage and are not intended for use beyond six (6) months.

All Motiva Flora® TE's require periodic, incremental inflation with sterile saline for injection until the desired tissue amount is developed. After the desired volume, the expander is surgically removed and replaced with a long-term breast implant in the same space as the tissue expander.

The study collects retrospective data on the use of the Motiva Flora TE, from patients who had a tissue expander-based-breast reconstruction using the Motiva Flora® TE since market introduction in May 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a tissue expander-based breast reconstruction with the Motiva Flora® TE .
* Patient has been informed correctly according to to the applicable national and local regulations.

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient has had a complete tissue-expander based breast reconstruction with the Motiva Flora® TE .
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Safety - adverse events | Until finalization of staged Breast reconstruction, approximately 6 months
  Cumulative incidence and causal relationship with the device of adverse events (AEs) reported by the surgeon. This includes known complications as listed in the IFU, as well as any other adverse events, seen as at least possibly related to the device according to the surgeon.
Safety - device deficiencies | Until finalization of staged Breast reconstruction, approximately 6 months
  Device-related complications include those resulting from any device failure, including those resulting in removal and/or replacement of the Motiva Flora® TE.
Performance - succesful implant of long-term breast implant | Until finalization of staged Breast reconstruction, approximately 6 months
  Successful tissue expander-based-breast reconstruction is measured by the fact that the second step of the staged procedure - the implantation of the long-term breast implant - could be performed or not as initially planned, as per surgeon judgement (Yes / No)
Performance - surgeon satisfaction | Until finalization of staged Breast reconstruction, approximately 6 months
  Surgeon's overall satisfaction with the results of the expansion according to the General Aesthetic Improvement Scale (GAIS), a 5-point Likert scale (1=very significant improvement, 2=significant improvement, 3=improvement, 4=no change and 5=decline) after the completion of the breast reconstruction (after the second surgery (long-term breast implant).

SECONDARY OUTCOMES:
Length of hospitalization | Until discharge from hospital after first surgery (Motiva Flora Tissue Expander), approximately 1-2 days
  Length of hospitalization is measured in number of days that the patient stays in hospital after surgery, starting from the day after surgery.
Surgical difficulties- 1st surgery (Motiva Flora TE implantation) | Intraoperative
  Possible difficulties during the during the 1st surgery, measured through the occurrence of:
  * device deficiencies / malfunctions
  * difficulties filling the Tissue expander with the Port Locator
Surgical difficulties - 2nd surgery (Long-term breast implant) | Intraoperative
  Possible difficulties during the 2nd surgery, measured through the occurrence of:
  o device deficiencies /malfunctions
Concomitant treatments - 1st surgery | Intraoperative
  Concomitant treatments during the 1st surgery is measured through the occurrence of:
  * Lipotransfer
  * Latissimus Dorsi Flap
Concomitant treatments - 2nd surgery | Intraoperative
  Concomitant treatments during the 2nd surgery is measured through the:
  * Use of Motiva Sizers
  * The occurrence of Lipotransfer

CONTACTS AND LOCATIONS:
Locations (2):
- Dr Filip Stillaert, Ghent, Belgium
- Fundacion Tejerina, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No